CLINICAL TRIAL: NCT02755532
Title: A Clinical and Pharmacokinetic Study to Evaluate the Influence of Two Bupivacaine Concentrations on Peak Plasma After Ultrasound-guided Axillary Brachial Plexus Block
Brief Title: Bupivacaine Pharmacokinetics in Ultrasound-guided Axillary Brachial Plexus Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Bupvacaine Pharmacokinetic
Record Dates: First submitted 2016-04-22; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Pharmacokinetics; Anesthetics, Local
Keywords: Pharmacokinetics; Bupivacaine; Axillary brachial plexus block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine 0,25% (Active Comparator): Routine surgical procedure monitoring with an electrocardiogram, sphygmomanometer, and pulse oximeter was performed. One experienced anesthesiologist performed an ultrasound guided axillary brachial plexus block (S Series, FUJIFILM Sonosite, Seattle, USA) with the patient in the supine position. Local anesthetic injection was performed on each nerve identified in this pathway (i.e., the radial nerve, the ulnar nerve, the median nerve, and the musculocutaneous nerve) In the group bupicavaine 0.25%, 10 ml of 0.25% bupivacaine was injected into each nerve, for a total of 40 ml per patient.
  Interventions: Drug: Bupivacaine 0,25%
- Bupivacaine 0,5% (Active Comparator): Routine surgical procedure monitoring with an electrocardiogram, sphygmomanometer, and pulse oximeter was performed. One experienced anesthesiologist performed an ultrasound guided axillary brachial plexus block (S Series, FUJIFILM Sonosite, Seattle, USA) with the patient in the supine position. Local anesthetic injection was performed on each nerve identified in this pathway (i.e., the radial nerve, the ulnar nerve, the median nerve, and the musculocutaneous nerve). In the group bupivacaine 0.5% , 5 ml of 0.5% bupivacaine was injected into each nerve, for a total of 20 ml per patient.
  Interventions: Drug: Bupivacaine 0,5%

INTERVENTIONS:
Drug: Bupivacaine 0,25% — Venous blood samples were collected prior to blocking , every 15 min during the first hour after completion of the blocking and every 30 min during the second hour after completion using an exclusive cannula. Then, 5 ml was drawn off and was stored in two EDTA tubes (BD, Franklin Lakes, NJ, USA). The EDTA tubes were centrifuged at 3,500xg for 10 min to obtain the blood plasma. This plasma was then stored in cryogenic tubes in a freezer at -80 °C until the time of the analysis. A high-performance liquid chromatography apparatus (Shimadzu, Kyoto, Japan) coupled to a Bruker mass spectrometer (MS), model Amazon (USA), with electrospray source ionization and a sequential mass spectrometry system (MS/MS) were used for the analysis. After obtaining the precursor ion, a fragment was obtained via a collision-induced dissociation process. The following molecular ions were selected: 289.0 m/z==>140.1 m/z. The methodology was validated according to the international FDA recommendations.
  Arms: Bupivacaine 0,25%
Drug: Bupivacaine 0,5% — Venous blood samples were collected prior to blocking , every 15 min during the first hour after completion of the blocking and every 30 min during the second hour after completion using an exclusive cannula. Then, 5 ml was drawn off and was stored in two EDTA tubes (BD, Franklin Lakes, NJ, USA). The EDTA tubes were centrifuged at 3,500xg for 10 min to obtain the blood plasma. This plasma was then stored in cryogenic tubes in a freezer at -80 °C until the time of the analysis. A high-performance liquid chromatography apparatus (Shimadzu, Kyoto, Japan) coupled to a Bruker mass spectrometer (MS), model Amazon (USA), with electrospray source ionization and a sequential mass spectrometry system (MS/MS) were used for the analysis. After obtaining the precursor ion, a fragment was obtained via a collision-induced dissociation process. The following molecular ions were selected: 289.0 m/z==>140.1 m/z. The methodology was validated according to the international FDA recommendations.
  Arms: Bupivacaine 0,5%

SUMMARY:
Introduction: The risk of systemic toxicity when using bupivacaine is a persistent problem, making its pharmacokinetic study crucial to the safety of regional anesthesia (RA). Little evidence exists regarding the effect of different concentrations of this drug on peak plasma levels. The present study compares two bupivacaine concentrations to establish how the concentration and exchange area affect the peak plasma level of this drug during axillary brachial plexus block. Latency and postoperative analgesia periods were also compared.

Methods: 32 patients were randomly assigned to two groups. In the 0.25% group, 10 ml of 0.25% bupivacaine was injected per nerve; in the 0.5% group, 5 ml of 0.5% bupivacaine was injected per nerve. Peripheral blood samples were collected every 15 min during the first hour and every 30 min during the second hour to establish serum level dosage. High-performance liquid chromatography coupled with mass spectrometry was used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* candidates for elective surgery of the distal forearm and hand for whom brachial plexus anesthesia and analgesia were indicated.
* physical status of I or II according to American Society of Anesthesiologists (ASA) criteria
* body mass index (BMI) of less than 35 kg/m2
* Signed the free and informed consent document.

Exclusion Criteria:

* cognitive impairment
* infection at the block puncture site
* coagulopathy
* history of bupivacaine allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Peak Venous Plasma level of bupivacaine. | 2 hours
  The aim of this study was to evaluate the difference in peak plasma levels obtained after ultrasound guided axillary brachial plexus block using two different bupivacaine concentrations to maintain the infused mass. Venous blood samples were collected prior to blocking , every 15 min during the first hour after completion of the blocking and every 30 min during the second hour after completion using an exclusive cannula. Then, 5 ml was drawn off and was stored in two EDTA tubes (BD, Franklin Lakes, NJ, USA). The EDTA tubes were centrifuged at 3,500xg for 10 min to obtain the blood plasma. This plasma was then stored in cryogenic tubes in a freezer at -80 °C until the time of the analysis. A high-performance liquid chromatography apparatus (Shimadzu, Kyoto, Japan) coupled to a Bruker mass spectrometer (MS), model Amazon (USA), with electrospray source ionization and a sequential mass spectrometry system (MS/MS) were used for the analysis.

SECONDARY OUTCOMES:
Latency - The latency period was defined as the time interval between time zero and the time when surgical anesthesia was obtained. | 30 minutes
  This evaluation occurred every 5 min until the 30th min after blocking. During this period, if surgical anesthesia was not obtained, then a complementary bupivacaine injection was administered distal to the axilla and the patient was excluded from the protocol. Surgical anesthesia was defined as a motor scale of 2 or lower; an absence of cold and pinprick sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo HC Ferraro, PhD, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulroy MF. Systemic toxicity and cardiotoxicity from local anesthetics: incidence and preventive measures. Reg Anesth Pain Med. 2002 Nov-Dec;27(6):556-61. doi: 10.1053/rapm.2002.37127. No abstract available. PMID 12430104
- [Background] Rosenberg PH, Veering BT, Urmey WF. Maximum recommended doses of local anesthetics: a multifactorial concept. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):564-75; discussion 524. doi: 10.1016/j.rapm.2004.08.003. PMID 15635516
- [Result] Liu SS, Ortolan S, Sandoval MV, Curren J, Fields KG, Memtsoudis SG, YaDeau JT. Cardiac Arrest and Seizures Caused by Local Anesthetic Systemic Toxicity After Peripheral Nerve Blocks: Should We Still Fear the Reaper? Reg Anesth Pain Med. 2016 Jan-Feb;41(1):5-21. doi: 10.1097/AAP.0000000000000329. No abstract available. PMID 26650424
- [Result] Vasques F, Behr AU, Weinberg G, Ori C, Di Gregorio G. A Review of Local Anesthetic Systemic Toxicity Cases Since Publication of the American Society of Regional Anesthesia Recommendations: To Whom It May Concern. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):698-705. doi: 10.1097/AAP.0000000000000320. PMID 26469367
- [Result] Dillane D, Finucane BT. Local anesthetic systemic toxicity. Can J Anaesth. 2010 Apr;57(4):368-80. doi: 10.1007/s12630-010-9275-7. Epub 2010 Feb 12. PMID 20151342
- [Result] Lee LA, Posner KL, Cheney FW, Caplan RA, Domino KB. Complications associated with eye blocks and peripheral nerve blocks: an american society of anesthesiologists closed claims analysis. Reg Anesth Pain Med. 2008 Sep-Oct;33(5):416-22. doi: 10.1016/j.rapm.2008.01.016. PMID 18774510
- [Result] Auroy Y, Narchi P, Messiah A, Litt L, Rouvier B, Samii K. Serious complications related to regional anesthesia: results of a prospective survey in France. Anesthesiology. 1997 Sep;87(3):479-86. doi: 10.1097/00000542-199709000-00005. PMID 9316950
- [Result] Takeda A, Ferraro LH, Rezende AH, Sadatsune EJ, Falcao LF, Tardelli MA. Minimum effective concentration of bupivacaine for axillary brachial plexus block guided by ultrasound. Braz J Anesthesiol. 2015 May-Jun;65(3):163-9. doi: 10.1016/j.bjane.2013.11.007. Epub 2015 Feb 16. PMID 25925026
- [Result] Cohen LS, Rosenthal JE, Horner DW Jr, Atkins JM, Matthews OA, Sarnoff SJ. Plasma levels of lidocaine after intramuscular administration. Am J Cardiol. 1972 Apr;29(4):520-3. doi: 10.1016/0002-9149(72)90442-0. No abstract available. PMID 5016830